CLINICAL TRIAL: NCT00620659
Title: Phase IIa, Randomized, Double-blind, Placebo-controlled, 3-period Crossover, Adaptive Dose Design, Clinical Trial to Evaluate Safety & Efficacy of MK0249 in Treating Refractory Excessive Daytime Sleepiness in Patients With Obstructive Sleep Apnea/Hypopnea Syndrome Appropriately Using nCPAP Therapy.
Brief Title: Treatment of Refractory Excessive Daytime Sleepiness in Patients With Obstructive Sleep Apnea/Hypopnea Syndrome (OSA/HS) Using Nasal Continuous Positive Airway Pressure (nCPAP) Therapy (0249-015)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0249-015; 2007_602
Record Dates: First submitted 2008-01-10; First posted 2008-02-21 (Estimated); Results first posted 2011-02-23 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-04

CONDITIONS: Sleep Apnea, Obstructive; Hypopnea Syndrome; Excessive Daytime Sleepiness
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- 1 (Experimental): Arm 1: Treatment period 1: MK0249; Treatment period 2: Placebo; Treatment period 3: modafinil
  Interventions: Drug: Comparator: MK0249; Drug: Comparator: placebo; Drug: Comparator: modafinil
- 2 (Experimental): Arm 2: Treatment period 1: Placebo; Treatment period 2: modafinil; Treatment period 3: MK0249
  Interventions: Drug: Comparator: MK0249; Drug: Comparator: placebo; Drug: Comparator: modafinil
- 3 (Experimental): Arm 3: Treatment period 1: modafinil; Treatment period 2: MK0249; Treatment period 3: Placebo
  Interventions: Drug: Comparator: MK0249; Drug: Comparator: placebo; Drug: Comparator: modafinil
- 4 (Experimental): Arm 4: Treatment period 1: MK0249; Treatment period 2: modafinil; Treatment period 3: Placebo
  Interventions: Drug: Comparator: MK0249; Drug: Comparator: placebo; Drug: Comparator: modafinil
- 5 (Experimental): Arm 5: Treatment period 1: Placebo; Treatment period 2: MK0249; Treatment period 3: modafinil
  Interventions: Drug: Comparator: MK0249; Drug: Comparator: placebo; Drug: Comparator: modafinil
- 6 (Experimental): Arm 6: Treatment period 1: modafinil; Treatment period 2: Placebo; Treatment period 3: MK0249
  Interventions: Drug: Comparator: MK0249; Drug: Comparator: placebo; Drug: Comparator: modafinil

INTERVENTIONS:
Drug: Comparator: MK0249 — Patients will be assigned to receive MK0249 film coated tablet (FCT). The doses of MK0249 that are included for possible investigation (depending upon an adaptive allocation process) are 3 mg, 5 mg, 8 mg, 10 mg, and 12 mg. Study medication will be taken for 14 days, during each of the 3 treatment periods, by mouth (po) once a day (qd).
Drug: Comparator: placebo — Placebo; Patients will be assigned to receive placebo, across 3 treatment periods. Study medication will be taken for 14 days, during each of the 3 treatment periods, po qd.
Drug: Comparator: modafinil — Patients will be assigned to receive modafinil 200mg oral compressed tablet (OCT), across 3 treatment periods. Study medication will be taken for 14 days, during each of the 3 treatment periods, po qd.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of MK0249 in treating refractory excessive daytime sleepiness (EDS) in patients with Obstructive Sleep Apnea/Hypopnea Syndrome (OSA/HS) using nasal continuous positive airway pressure (nCPAP) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female and is at least 18 years old and less than 65 years old
* Patient must have a diagnosis of Obstructive Sleep Apnea/Hypopnea Syndrome
* Patient has been using nCPAP treatment for at least 2 months prior to Visit 1
* Patient is willing to stay at a sleep laboratory for 4 full days and nights for observation and assessments
* Patient is willing to refrain from napping for the duration of the study

Exclusion Criteria:

* Patient is pregnant, breastfeeding, or planning to become pregnant within the next 4 months
* Patient is or has participated in a study with an investigational compound or device within 30 days of signing the informed consent
* Patient has had asthma-related visit to the emergency room or hospitalization within 6 months of Visit 1
* Patient has donated or received blood products within 8 weeks of signing consent or is planning on doing either for the duration of the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Herring WJ, Liu K, Hutzelmann J, Snavely D, Snyder E, Ceesay P, Lines C, Michelson D, Roth T. Alertness and psychomotor performance effects of the histamine-3 inverse agonist MK-0249 in obstructive sleep apnea patients on continuous positive airway pressure therapy with excessive daytime sleepiness: a randomized adaptive crossover study. Sleep Med. 2013 Oct;14(10):955-63. doi: 10.1016/j.sleep.2013.04.010. Epub 2013 Aug 3. PMID 23920422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The majority of patients were recruited from investigators' own databases at 24 sites in the United States. The primary therapy period was 13-Mar-2008 to 25-Feb-2009.
Pre-assignment Details: Participants maintained sleep and sleepiness diaries during a 7- to 10-day placebo run-in period. They used a nasal continuous positive airway pressure (nCPAP) device to monitor their CPAP use. At the end of the run-in period, participants stayed overnight at the clinic for nighttime polysomnography and if eligible, were randomized the next morning
Groups:
- MK0249/Placebo/Modafinil; Placebo/Modafinil/MK0249; Modafinil/MK0249/Placebo; MK0249/Modafinil/Placebo; Placebo/MK0249/Modafinil; Modafinil/Placebo/MK0249: Eligible participants were equally randomized to 1 of 6 treatment sequences: MK0249/Placebo/Modafinil, Placebo/Modafinil/MK0249, Modafinil/MK0249/Placebo, MK0249/Modafinil/Placebo, Placebo/MK0249/Modafinil, Modafinil/Placebo/MK0249. The dose of the MK0249 was determined according to a predefined adaptive algorithm. Treatment period was determined by the sequence to which the participant was randomized. Each treatment period was followed by a 7-day placebo washout period.
  MK0249 was provided as 1 mg and 5 mg tablets. Modafinil was provided as 100 mg tablets. Matching placebo tablets were provided for the MK0249 1 and 5 mg tablets and for the modafinil 100 mg tablet.
Period: Treatment Period 1
Arm/Group | MK0249/Placebo/Modafinil | Placebo/Modafinil/MK0249 | Modafinil/MK0249/Placebo | MK0249/Modafinil/Placebo | Placebo/MK0249/Modafinil | Modafinil/Placebo/MK0249
Started | 21 | 21 | 21 | 21 | 21 | 20
Completed | 18 | 21 | 20 | 18 (1 patient discontinued from MK0249, but continued in following periods, & completed the study) | 20 | 20
Not Completed | 3 | 0 | 1 | 3 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 3 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 1 | 0
Period: Placebo Washout Period 1
Arm/Group | MK0249/Placebo/Modafinil | Placebo/Modafinil/MK0249 | Modafinil/MK0249/Placebo | MK0249/Modafinil/Placebo | Placebo/MK0249/Modafinil | Modafinil/Placebo/MK0249
Started | 18 | 21 | 20 | 19 | 20 | 20
Completed | 18 | 21 | 20 | 18 | 20 | 20
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Period: Treatment Period 2
Arm/Group | MK0249/Placebo/Modafinil | Placebo/Modafinil/MK0249 | Modafinil/MK0249/Placebo | MK0249/Modafinil/Placebo | Placebo/MK0249/Modafinil | Modafinil/Placebo/MK0249
Started | 18 | 21 | 20 | 18 | 20 | 20
Completed | 18 | 18 | 19 | 18 | 15 | 20
Not Completed | 0 | 3 | 1 | 0 | 5 | 0
Not completed — Adverse Event | 0 | 3 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 3 | 0
Period: Placebo Washout Period 2
Arm/Group | MK0249/Placebo/Modafinil | Placebo/Modafinil/MK0249 | Modafinil/MK0249/Placebo | MK0249/Modafinil/Placebo | Placebo/MK0249/Modafinil | Modafinil/Placebo/MK0249
Started | 18 | 18 | 19 | 18 | 15 | 20
Completed | 16 | 18 | 19 | 18 | 15 | 20
Not Completed | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | MK0249/Placebo/Modafinil | Placebo/Modafinil/MK0249 | Modafinil/MK0249/Placebo | MK0249/Modafinil/Placebo | Placebo/MK0249/Modafinil | Modafinil/Placebo/MK0249
Started | 16 | 18 | 19 | 18 | 15 | 20
Completed | 16 | 16 | 19 | 17 | 15 | 20
Not Completed | 0 | 2 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All participants randomized in study
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 100
Race/Ethnicity, Customized [Number; unit: participants]
  White | 102
  Black or African American | 19
  American Indian or Alaska Native | 1
  Asian | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean of Average Maintenance of Wakefulness Test Early for The Mode Dose of MK0249 Versus Placebo
Description: The Maintenance of Wakefulness Test (MWT) is an objective assessment of sleepiness that measures the ability of a patient to remain awake. The primary endpoint was the mean of sleep latency (average of the first 4 MWTs which were at 0900, 1100, 1300, and 1500), where latency for each MWT was defined as the time to onset of the first 16 continuous seconds of any stage of sleep; if no sleep was observed according to these rules, then latency was defined as 30 minutes. The comparison was for the mode dose of MK0249 versus placebo.
Time Frame: At Week 2
Population: Full Analysis Set (FAS): The FAS population was a subset of all randomized patients with patients excluded for failure to receive at least one dose of study treatment or lack of endpoint data. Patients with at least one dose and endpoint in at least one treatment period were included in the FAS.
Measure: Least Squares Mean (Standard Error); unit: Minutes
Groups:
- Placebo: There were 116 participants who received placebo over 3 periods (42, 38, and 36 participants for Periods 1, 2, and 3 respectively).
- MK0249 Mode Dose: The Mode dose (the dose to which most patients were adaptively assigned) of MK0249 was 10 mg.
  There were 39 participants who received MK0249 10 mg (Mode Dose) over 3 periods (14, 12, and 13 participants for Periods 1, 2, and 3 respectively).
Arm/Group | Placebo | MK0249 Mode Dose
Number analyzed (Participants) | 116 | 39
Minutes | 12.79 (0.75) | 13.34 (1.09)
Statistical Analysis 1: Comparison: Placebo vs MK0249 Mode Dose; Test type: Superiority or Other; p = 0.615, Mixed Models Analysis; The mixed model included terms for period and treatment

2. Secondary Outcome: Mean of Average Maintenance of Wakefulness Test Early for the Mode Dose of MK0249 Versus Modafinil
Description: The Maintenance of Wakefulness Test (MWT) is an objective assessment of sleepiness that measures the ability of a patient to remain awake. The primary endpoint was the mean of sleep latency (average of the first 4 MWTs which were at 0900, 1100, 1300, and 1500), where latency for each MWT was defined as the time to onset of the first 16 continuous seconds of any stage of sleep; if no sleep was observed according to these rules, then latency was defined as 30 minutes. The comparison was for the mode dose of MK0249 versus modafinil.
Time Frame: At Week 2
Population: Full Analysis Set (FAS): The FAS population was a subset of all randomized patients with patients excluded for failure to receive at least one dose of study treatment or lack of an endpoint data. Patients with at least one dose and endpoint in at least one treatment period were included in the FAS.
Measure: Least Squares Mean (Standard Error); unit: Minutes
Groups:
- MK0249 Mode Dose: The Mode dose (the dose to which most patients were adaptively assigned) of MK0249 was 10 mg
  There were 39 participants who received MK0249 10 mg (Mode Dose) over 3 periods (14, 12, and 13 participants for Periods 1, 2, and 3 respectively).
- Modafinil 200 mg: There were 106 participants who received Modafinil 200 mg over 3 periods (40, 36, and 30 participants for Periods 1, 2, and 3 respectively).
Arm/Group | MK0249 Mode Dose | Modafinil 200 mg
Number analyzed (Participants) | 39 | 106
Minutes | 13.34 (1.09) | 17.45 (0.74)
Statistical Analysis 1: Comparison: MK0249 Mode Dose vs Modafinil 200 mg; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 1.5 minutes. If the lower bound of the one-sided 95% confidence interval for MK0249 minus modafinil 200 mg was greater than -1.5 minutes, non-inferiority would be established; Difference in Least Squares Mean = -4.11, 90% CI 2-sided [-5.92 to -2.30]

3. Secondary Outcome: Mean of Average Maintenance of Wakefulness Test Early for Top 2 Doses Pooled of MK0249 Versus Modafinil
Description: The Maintenance of Wakefulness Test (MWT) is an objective assessment of sleepiness that measures the ability of a patient to remain awake. The primary endpoint was the mean of sleep latency (average of the first 4 MWTs which were at 0900, 1100, 1300, and 1500), where latency for each MWT was defined as the time to onset of the first 16 continuous seconds of any stage of sleep; if no sleep was observed according to these rules, then latency was defined as 30 minutes. The comparison was for the top 2 doses pooled of MK0249 versus modafinil.
Time Frame: At Week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Minutes
Groups:
- MK0249 Top 2 Doses Pooled: The top 2 doses (the two doses to which most patients were adaptively assigned) were 10 mg and 12 mg.
  There were 74 participants who received MK0249 10 and 12 mg over 3 periods (25, 22, and 27 participants for Periods 1, 2, and 3 respectively).
Arm/Group | MK0249 Top 2 Doses Pooled | Modafinil 200 mg
Number analyzed (Participants) | 74 | 106
Minutes | 13.64 (0.85) | 17.45 (0.74)
Statistical Analysis 1: Comparison: MK0249 Top 2 Doses Pooled vs Modafinil 200 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in Least Squares Mean = -3.80, 90% CI 2-sided [-5.23 to -2.38]

4. Secondary Outcome: Clinical Global Impressions Scale of Severity Score as it Relates to Excessive Daytime Sleepiness (CGIS-EDS) for the Mode Dose of MK0249 Versus Placebo
Description: Clinical Global Impressions Scale of Severity (CGI-S) is a subscale of the CGI which is a standard psychometric scale used to demonstrate changes and improvements in illness. CGI-S consists of a 7-point scale rated from 1 to 7. The investigator or sponsor-approved clinician judged how ill the patient was with respect to Excessive Daytime Sleepiness (EDS) at the time of the CGI-S rating (CGIS-EDS), with higher scores indicating more severe illness.
Time Frame: At Week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MK0249 Mode Dose
Number analyzed (Participants) | 116 | 39
units on a scale | 3.76 (0.11) | 3.43 (0.18)
Statistical Analysis 1: Comparison: Placebo vs MK0249 Mode Dose; Test type: Superiority or Other; p = 0.079, Mixed Models Analysis; The mixed model included terms for period and treatment

5. Secondary Outcome: Epworth Sleepiness Scale (ESS) Score for the Mode Dose of MK0249 Versus Placebo
Description: The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire that provides subjective reports that equate with sleep propensity, not with 'subjective sleepiness'. Having a high sleep propensity means having a history of dozing in situations that have a relatively low soporific nature, in which normal subjects seldom doze. The ESS consists of eight items, which are rated from 0 ("would never dose") to 3 ("high chance of dozing"). The ESS score is the total score of the 8 individual items; this total score ranges from 0 to 24 (higher total score is worse).
Time Frame: At Week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MK0249 Mode Dose
Number analyzed (Participants) | 115 | 40
units on a scale | 12.81 (0.43) | 10.83 (0.65)
Statistical Analysis 1: Comparison: Placebo vs MK0249 Mode Dose; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; The mixed model included terms for period and treatment

ADVERSE EVENTS:
Time Frame: Patients reported adverse experiences starting from the Screening Visit up until 14 days after the last dose of study drug.
Description: Patients reported AEs at each visit, and the occurrence of serious adverse experiences was assessed during a telephone contact fourteen days after the last dose of study drug.
Groups:
- Placebo: Matching placebo tablets were provided for the MK0249 1 and 5 mg tablets and for the modafinil 100 mg tablet.
- MK0249 5 mg; MK0249 8 mg; MK0249 10 mg; MK0249 12 mg: MK0249 was provided as 1 mg and 5 mg tablets.
- Modafinil: Modafinil was provided as 100 mg tablets.
Arm/Group | Placebo | MK0249 5 mg | MK0249 8 mg | MK0249 10 mg | MK0249 12 mg | Modafinil
Serious Adverse Events (participants affected / at risk) | 2/117 | 0/10 | 0/25 | 0/46 | 0/39 | 0/111
Other Adverse Events (participants affected / at risk) | 41/117 | 6/10 | 7/25 | 16/46 | 25/39 | 38/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=117) | MK0249 5 mg (N=10) | MK0249 8 mg (N=25) | MK0249 10 mg (N=46) | MK0249 12 mg (N=39) | Modafinil (N=111)
Acute pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymph node abscess (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=117) | MK0249 5 mg (N=10) | MK0249 8 mg (N=25) | MK0249 10 mg (N=46) | MK0249 12 mg (N=39) | Modafinil (N=111)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ear buzzing (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Scleral haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Subconjunctival ecchymosis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Burping (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Gastric pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Malodorous burping (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 2
Stomach ache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomach fullness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Upset stomach (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 3
Application site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Chest pressure (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest tightness (General disorders) | 1 | 0 | 0 | 1 | 0 | 1
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Foot oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hand swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hangover (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Implant site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Increased thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 1 | 1 | 2
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Liver fatty (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cold (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 1
Cold sores (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cold symptoms (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Head cold (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pinkeye (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sinus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Yeast infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Back strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Contusion of upper arm (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Device induced injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Laceration of foot (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Lateral epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Leg injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Pulled muscle (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Shoulder sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood sugar increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Creatine phosphokinase increased (Investigations) | 1 | 1 | 1 | 0 | 1 | 2
Glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Glucose urine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Urine calcium oxalate crystal present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Appetite lost (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back ache (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Knee pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Low back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Muscle ache (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pain in leg (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sore back (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Attention concentration difficulty (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Concentration impaired (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Head pressure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 7 | 1 | 0 | 2 | 4 | 12
Headache dull (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypnagogic myoclonus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lightheadedness (Nervous system disorders) | 2 | 0 | 0 | 1 | 1 | 1
Nocturnal headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus pressure (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Taste metallic (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tingling feet/hands (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 3 | 3 | 3 | 1
Bad dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dreaming excessive (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 3 | 7 | 11 | 2
Middle insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mood change (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 2
Nocturnal awakening (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Sleep maintenance insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sleep talking (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Teeth clenching (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vivid dreams (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 0
Kidney stone (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ejaculation delayed (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Breath shortness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasal sinus discharge (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasal stuffiness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Clamminess (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diaphoresis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hives (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ingrown toe nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Localised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Feeling of hot flushes (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Generalised flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.